CLINICAL TRIAL: NCT04316442
Title: A Phase 1b/2a, Open-Label, Dose-Escalation Study of the Safety and Efficacy of an Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With Relapsed or Refractory Systemic AL Amyloidosis
Brief Title: Study of the Safety and Efficacy of STI-6129 in Patients With Relapsed or Refractory Systemic AL Amyloidosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STI-6129-001
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Light Chain (AL) Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-6129 infusion (Experimental): Intravenous infusion to be given with prophylaxis for infusion reactions if necessary.
  Interventions: Biological: STI-6129

INTERVENTIONS:
Biological: STI-6129 — Four cycles of intravenous infusion of STI-6129 will be given (one infusion every four weeks).
  Other Names: anti-CD38-Duostatin 5.2 antibody-drug conjugate (ADC)

SUMMARY:
The STI-6129-001 study is a three-stage, multicenter, open-label, dose-finding, phase 1b/2a trial. It is designed primarily to identify the recommended phase 2 dose (RP2D) of STI-6129 by assessing the safety, preliminary efficacy and pharmacokinetics of this anti-CD38-Duostatin 5.2 antibody-drug conjugate (ADC) for the treatment of relapsed or refractory systemic AL amyloidosis.

The patients that will be treated with STI-6129 in this trial are relapsed or refractory systemic AL amyloidosis patients who have received prior lines of treatment.

DETAILED DESCRIPTION:
This study is composed of three dosing plan stages. The initial stage of this trial is the dose-escalation stage. A modified dose-escalation 3+3 design will be utilized to identify a safe maximum tolerated dose (MTD) of STI-6129 in patients with relapsed or refractory systemic AL amyloidosis. After identification of the MTD, or the finding that the last dosing cohort is tolerated well (i.e., the maximum practical dose [MPD]), 12 patients will be enrolled to receive STI-6129 treatment at the MTD/MPD level to collect pharmacokinetic data ( the pharmacokinetic (PK) stage) to model a treatment schedule that achieves a stable effective serum concentration. Results from the dose-escalation stage and the pharmacokinetic stage will be analyzed to develop a treatment dose/schedule for treating 30 additional patients enrolled in the expansion stage.

Each patient enrolled will receive up to three 4-week cycles of STI-6129, unless a longer intermission is required. After the treatment period, patients will be monitored for up to a year.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AL amyloidosis by tissue biopsy of an involved organ, or a surrogate site such as abdominal fat demonstrating amyloid deposition by mass spectrometry
* The presence of a monoclonal light chain protein in serum
* Relapsed or refractory AL amyloidosis is defined as patients who have received ≥ 2 lines of treatment. Patients must have received at least one proteasome inhibitor during their prior therapy. Patients who have received prior daratumumab treatment or prior stem cell transplantation remain eligible. Patients may have relapsed with disease progression or have been refractory to their last prior line of treatment. Progression of disease that develops > 60 days after the last dose of a treatment regimen in a patient who achieved at least a partial response (PR) defines a relapse. Refractory systemic AL amyloidosis is defined as the development of disease progression during therapy with an anti-AL amyloidosis treatment regimen or within 60 days of the last dose of an anti-AL amyloidosis treatment regimen or the achievement of less than a PR after ≥ 2 cycles
* Measurable disease defined as the finding by serum-free light chain (FLC) assay that the difference between the involved and uninvolved FLC (dFLC) is ≥ 50 mg/L
* Pulse oximetry ≥ 92% on room air
* ECOG performance status of 0, 1, or 2
* Willing to comply with the study schedule and all other protocol requirements
* Females of childbearing potential (FCBP) must have 2 negative pregnancy tests prior to treatment. All heterosexually active FCBP and all heterosexually active male patients must agree to use effective methods of birth control throughout the study

Exclusion Criteria:

* Isolated vascular amyloid in a bone marrow biopsy or a plasmacytoma specimen or isolated soft tissue involvement (localized AL amyloidosis)
* Presence of non-AL amyloidosis
* A diagnosis of multiple myeloma
* A diagnosis of other malignancies if the malignancy has required therapy within the last 3 years or is not in complete remission. Exceptions are non-metastatic basal cell or squamous cell carcinomas of the skin or prostate cancer that does not require treatment
* Treatment with an allogeneic hematopoietic stem cell transplantation (HSCT) within 6 months prior to the planned infusion of STI-6129, or active graft-versus-host disease (GVHD) following the allogeneic transplant, or a requirement for currently receiving immunosuppressive therapy following the allogeneic transplant
* Revised Mayo Clinic AL amyloidosis stage > 3
* New York Heart Association (NYHA) class > 2
* Left ventricular ejection fraction (LVEF) < 40%
* Patients with mean left ventricular wall thickness ≥ 12 mm and/or intraventricular septal thickness > 25 mm by echocardiogram in the absence of hypertension or valvular heart disease
* Patients with NT-proBNP ≥ 1800 ng/L or BNP ≥ 400 ng/L, or cTNT ≥ 0.025 μg/L will be excluded in the dose-escalation stage of the study and can only be included in the PK and expansion stages after evaluation by cardiology and discussion with the principle investigator regarding the risk associated with the treatment
* Abnormal baseline hematological laboratory results at Screening:

  * Hemoglobin < 8.0 g/dL
  * Platelet count < 50,000/μL
  * Absolute neutrophil count (ANC) < 1000/μL
* Abnormal baseline chemistry laboratory results at Screening:

  * Serum creatinine ≥ 2.0 mg/dL or estimated creatinine clearance < 60 mL/min (using the Cockcroft-Gault equation)
  * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x the upper limit of normal (ULN) or serum total bilirubin > 1.5x ULN (except for patients in whom hyperbilirubinemia is attributed to Gilbert's Syndrome)
* INR or aPTT > 1.5x ULN within 1 week prior to the infusion of STI-6129, unless on a stable dose of an anticoagulant
* Pregnant or breastfeeding
* Active bacterial, viral, or fungal infection within 72 hours of the infusion of STI-6129; patients with ongoing use of prophylactic antibiotics, antifungal agents, or antiviral agents remain eligible as long as there is no evidence of active infection
* Have human immunodeficiency virus (HIV) infection, human T-cell leukemia virus type 1 (HTLV1) infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or are at risk for HBV reactivation (at risk for HBV reactivation is defined as being HBs antigen positive, or anti-HBc-antibody positive), or are positive for HBV deoxyribonucleic acid (DNA). HCV ribonucleic acid (RNA) must be undetectable by laboratory test
* QTcF > 470 msec on a baseline ECG
* Any condition including the presence of laboratory abnormalities that places the patient at unacceptable risk if the patient was to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of STI-6129 in AL amyloidosis patients | Baseline through study completion at up to 14 months
  Types, frequencies, and severities of adverse events (AEs) and the relationships of AEs to study drug; includes serious adverse events (SAEs), neurotoxicity, dose-limiting toxicities (DLTs), and laboratory abnormalities

SECONDARY OUTCOMES:
Overall hematological response rate according to the 2012 Consensus Round Table response criteria | Baseline through study completion at up to 14 months
  Proportion of subjects with Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), No Response (NR) and Progressive Disease (PD)
Organ response rates (cardiac, renal, hepatic, peripheral nervous system) according to the 2012 Consensus Round Table response criteria | Baseline through study completion at up to 14 months
  Organ response rates (cardiac, renal, hepatic, peripheral nervous system) according to the 2012 Consensus Round Table response criteria
Correlation of treatment response (organ responses and hematological response) with disease severity based on the 2012 revised Mayo Clinic staging system for AL amyloidosis | Baseline through study completion at up to 14 months
  Correlation of treatment response (organ responses and hematological response) with disease severity based on the 2012 revised Mayo Clinic staging system for AL amyloidosis
Plasma levels of the total antibody plus conjugated toxin (STI-6129) and the free toxin (Duostatin 5.2) | Day 1 to day 63
  Plasma levels of the total antibody plus conjugated toxin (STI-6129) and the free toxin (Duostatin 5.2) by ELISA and mass spectrophotometry assays, respectively, at pre-dose and various time points post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center; Michael Rosenzweig, MD, Principal Investigator — City of Hope National Medical Center; Jeffrey Zonder, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute Wertz Clinic; Anita D'Souza, MD, Principal Investigator — Froedtert Hospital & the Medical College of Wisconsin
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Boston Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute Wertz Clinic, Detroit, Michigan
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No